CLINICAL TRIAL: NCT05455827
Title: Using Functional MRI Neurofeedback to Modulate Self-blame in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton & Sussex Medical School (Other)
Responsible Party: Principal Investigator, James Stone, Prinicipal Investigator, Brighton & Sussex Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: US_FMRI_NF_JMS1
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Depression
Keywords: Neurofeedback; fMRI; MDD
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A (Experimental): Enhancing condition differences between guilt and indignation BOLD activations of subgenual anterior cingulate cortex.
  Interventions: Other: fMRI neurofeedback (A)
- Intervention B (Active Comparator): Minimising condition differences between guilt and indignation BOLD activations of subgenual anterior cingulate cortex.
  Interventions: Other: fMRI neurofeedback (B)

INTERVENTIONS:
Other: fMRI neurofeedback (A) — Participants will be shown feedback about the BOLD activation within the subgenual anterior cingulate cortex to enhance differences between the self-blame and other-blame conditions
  Arms: Intervention A
Other: fMRI neurofeedback (B) — Participants will be shown feedback about the BOLD activation within the subgenual anterior cingulate cortex to minimise differences between the self-blame and other-blame conditions
  Arms: Intervention B

SUMMARY:
To determine the feasibility of functional MRI neurofeedback in reducing overgeneralised self-blame in patients with depression

DETAILED DESCRIPTION:
Background

Low self-worth has been identified as a core cognitive symptom of major depressive disorder. Interestingly, brain activity markers of low self-worth remain somewhat present even after symptomatic remission. Consequently, these brain signatures could potentially be used to predict relapse. Low self-worth is thought to be underpinned by overgeneralised self-blame, where an individual shows a bias towards emotions of guilt and worthlessness, as opposed to indignation (the blame of others). Unfortunately, many current treatments for MDD do not address low self-worth specifically, and this might result in patients not responding as well as they could. Therefore, it would be beneficial to further investigate which areas of the brain are responsible for regulating excessive self-blaming emotions, in order to develop more targeted therapies and tools for managing the disorder.

In this study, the investigators will use a brain-scanning technique called 'fMRI neurofeedback' with a group of (current) MDD patients to try to change brain activity, in a specific region associated with self-blaming emotions, towards a healthier pattern. To clarify, in fMRI the brain is scanned to provide functional data (i.e. which brain regions are more / less active during a certain condition or task). fMRI with neurofeedback, however, is a relatively recent approach, which aims to show patients their fMRI data in real-time, while they are still in the scanner. Of course, this is presented to the patient in a simplified and abstracted form, such as a thermometer reading, whereby the thermometer level changes based on changes in brain activity. In this way, patients can learn to modulate their own brain activity in real-time towards healthier or more optimal patterns.

Previous neurofeedback studies of self-blame have instead used a target that is based on the functional connectivity dynamics between the right superior anterior temporal lobe (ATL) and the subgenual cingulate cortex (SCC). Whilst ATL-SCC connectivity has proven to be a good biomarker of self-blame, results concerning which direction is therapeutic (i.e. higher or lower connectivity) have been conflicting. Even when looking at SCC activity in isolation, the results are in opposition: some studies have suggested that minimizing differences in SCC activity between self-blame and other-blame conditions is beneficial, whereas recent unpublished findings suggest the reverse to be true (Fennema et al.). Consequently, there is a clear need to clarify which training direction is most therapeutic for MDD patients before the field rushes ahead. Conceivably, it is more straightforward to do this for the SCC in isolation, rather than for a pair of regions or a wider network, given that there will be a stronger and more reproducible response. Therefore, the current study will use activity in the SCC region as the sole neurofeedback target, in the interest of safety, simplicity and clarity.

The investigators will investigate two different neurofeedback designs, involving the SCC, in two different MDD patient groups to test which is most therapeutic for MDD patients. One group will be encouraged to increase differences in SCC activity between guilt and indignation conditions, and the other group will be encouraged to minimize differences. Both of these training directions, while different to each other, represent activation patterns that have been observed in healthy control populations (Zahn et al., 2009; Green et al., 2012; Fennema et al. (unpublished)). Therefore, the investigators are confident that neither intervention will incur any significant worsening of symptoms. Instead, the investigators hypothesize that both groups will be able to self-modulate activity in this region towards the target level and that, in at least one of the groups, this will be associated with improvements in self-worth ratings. As this study includes patients with current depression, rather than remitted depression, findings from this study will be more relevant to the ultimate target patient population.

In summary, this clinical proof-of-concept study addresses important gaps in our understanding of the field, and continues its overarching narrative closer towards decisions about clinical feasibility and implementation.

Aims

The investigators will harness the SCC, a brain region with an established role in regulating self-blame, as the target for a new fMRI neurofeedback trial of self-blame. This trial will include patients with current MDD. Both Intervention groups (A and B) will attempt to self-modulate their real-time fMRI blood oxygen level-dependent (BOLD) signal at the SCC which will be viewed as a thermometer-like reading. In the Intervention A group, participants will be encouraged to increase the differences in SCC BOLD activity between guilt and indignation conditions. In the Intervention B group, participants will be encouraged to minimize SCC BOLD activity between these conditions.

The guilt and indignation conditions refer to time points during the neurofeedback session when participants will be asked to experience emotions of guilt or indignation (at the same time as they try to raise the thermometer level) to determine whether brain activity changes are specific for emotions of self-blame or the blame of others. Implementation of the neurofeedback will be done through FRIEND software.

The investigators hypothesize that both groups will be able to self-modulate their neural signature towards the target level and that, in at least one of the intervention groups, this will correlate with improved ratings of self-worth at the clinical level.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent. Participants will be asked to complete consent before trial begins
* Understanding of verbal and written information given in English
* Online access
* Aged 18 or over
* Male or female
* Clinical diagnosis of MDD, with the following characteristics:

  * Meets Diagnostic and Statistical Manual V (DSM-V) criteria for MDD
  * Experience of a previous major depressive episode (MDE) lasting at least two months (evidence of recurrent depression)
  * Patients must have stable symptoms, lasting at least six weeks before experimental group randomisation
  * Exhibiting at least partial treatment resistance, evidenced by insufficient response to at least one psychological intervention or antidepressant intervention
  * Current use of antidepressants is not basis for exclusion, but patients must be on a stable dose for at least six weeks without improvement before the study start, and must remain at this dose throughout the study

Exclusion Criteria:

* Standard reasons for being unable to undergo MRI (e.g. metal implants)
* Impairments of vision or hearing which cannot be corrected for during the treatment sessions
* Pregnant or breastfeeding
* History of manic or hypomanic episodes, or schizophreniform or schizophrenia symptoms, or substance abuse
* History of violent behaviour or aggressive impulses
* History of neurological disorders such as seizures, loss of consciousness following brain injury or medical disorders affecting brain function, blood flow or metabolism
* History of learning disabilities, major medical, developmental or relevant other axis-I disorders
* Prior specialist diagnosis of attention deficit hyperactivity disorder (ADHD), antisocial or borderline personality disorder
* Significant impairment of psychosocial functioning before the last MDE indicating the possibility of a comorbid personality disorder or autism spectrum disorder
* Current intake of benzodiazepines, GABAergic or benzodiazepine receptor agonists
* Current recreational drug use
* Having MDD with the following characteristics:

  * Presenting with greater than 'low-risk' suicidality, violence or current self-harming behaviour
  * Experiencing a current MDE lasting more than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
BOLD activity in subgenual anterior cingulate | Acquired during the procedure
  Determine whether participants are able to modulate their anterior cingulate BOLD activity in keeping with the neurofeedback

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Clinician rated depression scale Score range: 0-60 Interpretation: higher score = worse outcome
Rosenberg self-esteem scale | 2 weeks before and at weeks 2, 4 and 6 after the fMRI neurofeedback session
  Self-esteem scale Score range: 10-40 Interpretation: higher score = better outcome
Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR-16) | 2 weeks before and at weeks 2, 4 and 6 after the fMRI neurofeedback session
  Self-rated depression scale Score range: 0-27 Interpretation: higher score = worse outcome
Generalised Anxiety Disorder Assessment (GAD-7) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Self-rated anxiety scale Score range: 0-21 Interpretation: higher score = worse outcome
Positive and Negative Affect Schedule (PANAS) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Self-rated measure of both positive and negative affect. Score range (Positive Affect): 10-50 Interpretation (Positive Affect): higher score = better outcome Score range (Negative Affect): 10-50 Interpretation (Negative Affect): higher score = worse outcome
Longitudinal Interval Follow-Up Evaluation (LIFE) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Score range (Psychiatric Status Rating): 0-6 Interpretation (Psychiatric Status Rating): higher score = worse outcome Score range (Psychosocial Functioning): 0-6 or 0-8 Interpretation (Psychosocial Functioning): higher score = worse outcome Score range (Global Assessment of Functioning): 0-100 Interpretation (Global Assessment of Functioning): higher score = better outcome Score range (Social and Occupational Functioning Assessment Scale): 0-100 Interpretation (Social and Occupational Functioning Assessment Scale): higher score = better outcome
Personal Style Inventory (PSI-II) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Score range (Sociotropy): 24-144 Interpretation (Sociotropy): n/a Score range (Autonomy): 24-144 Interpretation (Autonomy): n/a
Association for Methodology and Documentation in Psychiatry (AMDP) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Score range: 0-75 Interpretation: higher score = worse outcome
Value-related Moral Sentiment Task (VMST) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Value-related Moral Sentiment Task
Conceptual Social Knowledge Differentiation Task (CSKD) | 2 weeks before and 2 weeks after fMRI neurofeedback intervention
  Conceptual Social Knowledge Differentiation Task

CONTACTS AND LOCATIONS:
Locations (1):
- CISC, Brighton and Sussex Medical School., Brighton, East Sussex, United Kingdom